CLINICAL TRIAL: NCT04315038
Title: Metabolomics Profiling and Biomarker Research of Human Cerebrospinal Fluid in Aging Process and Age-related Neurodegenerative Diseases
Brief Title: Metabolomics Profiling Research of Human Cerebrospinal Fluid in Aging Process
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801931A
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-01

CONDITIONS: Aging; Metabolites; Neurodegenerative Diseases
Keywords: Aging; cerebrospinal fluid; metabolomics
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF samples will be stored in aliquots at -80 °C before analysis. The sample will be analyzed using hydrogen-1 nuclear magnetic resonance (1H-NMR) and lipid chromatography-mass spectrometry (LC-MS) in the Metabolomic Core Laboratory at Chang Gung Memorial Hospital or Chang Gung University. Demographic data including age, gender, body weight, blood pressure and past medical data will be investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Spinal anesthesia
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Plan to enroll 200 health volunteers and 40 neurodegenerative diseases patients with received spinal anesthesia. Blood will be collected at time point of pre-anesthesia 10 minutes and CSF samples will be collected at time point during spinal anesthesia induction. Blood will be collected, drawn into EDTA-coated tube.

SUMMARY:
Perform quantitative metabolomics on human cerebrospinal fluid (CSF) samples and establish the first human CSF Metabolome Database of aging process in Taiwan.

DETAILED DESCRIPTION:
Metabolomics is new science based on metabolite profiles in biofluids and tissues, which under bioinformatics approaches and analyses could help to characterize metabolomic status of CSF in aging process. In this prospective study, the investigators plan to enroll 200 health volunteers and 40 neurodegenerative diseases patients with received operation under spinal anesthesia. Blood and CSF samples will be analyzed using hydrogen-1 nuclear magnetic resonance (1H-NMR) and lipid chromatography-mass spectrometry (LC-MS).

ELIGIBILITY:
Inclusion Criteria:

Aging groups:

1. . Above 20 years.
2. . No history of central nerve system injury and neurologic illness
3. . ASA≦II
4. . Written informed consent from the patient

Aged-related neurodegenerative diseases group:

1. . Above 60 years of age
2. . Medical record proved the history of Parkinsonism or Alzheimer disease
3. . ASA≦III
4. . Written informed consent from the patient or guardian by statute.

Exclusion Criteria:

1. patient refuses to sign informed consent
2. patients with coagulopathy, systemic infective disease and severe liver and renal function impairment
3. patients with spine or brain tumor and CNS disease
4. the presence of severe and/or uncontrolled and/or unstable medical disease within 12 months prior to study (e.g. acute pancreatitis, stroke, liver cirrhosis, congestive heart failure, and systemic immune disorder etc
5. Concurrent participation or planning to participate in another interventional clinical trial (Concurrent participation in an observational trial allowed)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with received spinal anesthesia and had written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Exam metabolic profiles of CSF in aging process and age-related neurodegenerative diseases | An average of 1 year
  Metabolites analysis of CSF will be investigated by NMR, LC-MS. Peak lists of all NMR and LC/MS/MS spectra will be searched against the database through a web server for metabolomic data analysis and further establish the CSF Metabolome Database.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan